CLINICAL TRIAL: NCT02557854
Title: HIFU Hyperthermia With Liposomal Doxorubicin (DOXIL) for Relapsed or Refractory Pediatric and Young Adult Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Theodore Laetsch (Other)
Responsible Party: Sponsor-Investigator, Theodore Laetsch, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTSW-HIFU-001
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Rhabdomyosarcoma; Neuroblastoma; Sarcoma; Sarcoma, Ewing; Osteosarcoma; Desmoid
MeSH Terms: conditions — Rhabdomyosarcoma; Neuroblastoma; Sarcoma; Sarcoma, Ewing; Osteosarcoma; Desmoid Tumors | interventions — liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxil + MR-HIFU Hyperthermia (Experimental): Liposomal doxorubicin (Doxil) 50mg IV every 4 weeks followed by Magnetic Resonance High Intensity Focused Ultrasound hyperthermia (MR-HIFU) with Philips Sonalleve System to 42C for 30 minutes every 4 weeks
  Interventions: Drug: Doxorubicin HCl liposomal injection; Device: Philips Sonalleve MR-HIFU Hyperthermia

INTERVENTIONS:
Drug: Doxorubicin HCl liposomal injection — 50mg IV every 4 weeks
  Other Names: Doxil
Device: Philips Sonalleve MR-HIFU Hyperthermia — Hyperthermia to 42C for 30 minutes every 4 weeks

SUMMARY:
The purpose of this study is to determine whether Doxil (liposomal doxorubicin) given prior to MR-HIFU Hyperthermia is safe for the treatment of pediatric and young adult patients with recurrent and refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-40 years
* Histologically confirmed malignant extra-cranial solid tumor or demoid fibromatosis
* The subject's tumor must have relapsed after or failed to respond to frontline therapy and there must be no other known curative therapies available. Patients with desmoid fibromatosis must have relapsed after or failed to respond to at least one prior line of therapy, and in the opinion of the treating physician surgical resection of the tumor must not be possible without an amputation or other surgery predicted to result in an unacceptable functional deficit.
* Subject must have a life expectancy of > 8 weeks
* Karnofsky performance status > 50% for patients >16 years of age, or Lansky performance status > 50% for patients < 16 years of age.
* The subject must have at least 1 measurable target lesion >10mm in longest dimension that is in an anatomic location treatable by MR-HIFU. Note that for this study, lesions in bone WILL be considered measurable provided they meet the other criteria by RECIST and are confirmed to be metabolically active on baseline studies by either MIBG uptake (for neuroblastomas) or PET avidity. Target lesions should be located so that they can be adequately heated by a hyperthermia treatment cell with a diameter of up to 58 mm, centered at a depth of 35 to 80 mm from the skin. There should be no staples, implants, extensive scarring, or other highly ultrasound absorbing or reflecting tissue in the expected beam path. For the first 5 patients enrolled on this study only, the lesion must be located in the extremities or pelvis to be considered treatable by MR-HIFU.
* The subject must have recovered from the acute toxic effects of all prior therapy with the exception of alopecia. The following time must have elapsed from the last dose of the following medications to study enrollment:

  * myelosuppressive chemotherapy 14 days
  * hematopoetic growth factors 7 days (14 days for Neulasta)
  * biologic agent 7 days
  * monoclonal antibody 3 half-lives
  * immunotherapy (ie tumor vaccines) 42 days
  * palliative small port XRT 14 days
  * substantial bone marrow XRT 6 weeks
  * stem cell transplant or infusion without TBI 12 weeks
  * total body irradiation (TBI) 24 weeks
* Adequate organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1,000/mcL
  * platelets ≥ 75,000/mcl (without transfusion for 7 days)
  * hemoglobin > 8g/dL (may receive transfusions)
  * total bilirubin < 1.5 mg/dL
  * ALT(SPGT) < 225 U/L (45 U/L defined as ULN)
  * creatinine clearance or radioisotope GFR > 70 mL/min/1.73m2 OR a serum creatinine (mg/dL) less than or equal to the following:
  * Age (yrs)-----Male (mg/dL)-----Female (mg/dL)
  * 1-1.99----------0.6------------------0.6
  * 2-5.99----------0.8------------------0.8
  * 6-9.99----------1--------------------1
  * 10-12.99------1.2------------------1.2
  * 13-15.99------1.5------------------1.4
  * >16-------------1.7------------------1.4
* Adequate cardiac function defined as an ejection fraction > 50% or shortening fraction > 27%
* Cumulative lifetime anthracycline dose of < 450mg/m2
* Females and males of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A male of child-bearing potential is any male (regardless of sexual orientation, having undergone a vasectomy, or remaining celibate by choice) who has attained Tanner stage III or greater sexual development. A female of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has undergone menarche OR is > 13 years of age
* Females of child-bearing potential must have a negative serum pregnancy test within 7 days of treatment.
* Signed written informed consent must be obtained prior to any study procedures.

Exclusion Criteria:

* Subjects may not be receiving any other investigational agents or anticancer therapies.
* Subjects with known active brain metastases will be excluded from this clinical trial. Patients with brain metastases that have been treated and stable for > 30 days following treatment will be eligible.
* Subjects who have received prior Doxil and progressed on this therapy are not eligible, but subjects may have received prior doxorubicin.
* Subjects with a history of tumor progression within 30 days of anthracycline administration are not eligible. However, subjects who have previously received an anthracycline and subsequently relapse greater than 30 days after their most recent prior dose of anthracycline will be eligible.
* History of allergic reactions attributed to doxorubicin or Doxil
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Subjects with a contraindication to MR-HIFU
* Subjects with conditions that carry high anesthetic risk in the opinion of the treating anesthesiologist are not eligible (i.e. subjects with significant airway compression by tumor or craniofacial abnormalities)

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-03-16 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) during cycle 1 of therapy with MR-HIFU hyperthermia directed liposomal doxorubicin | 4 weeks
  Dose limiting toxicities are generally CTCAE v4.03 grade 3-5 toxicities with specific exceptions detailed in the protocol.

SECONDARY OUTCOMES:
Terminal half-life (T1/2) of Doxil when delivered with MR-HIFU hyperthermia | 48 hours following first dose
Volume of distribution (L/m2) of Doxil when delivered with MR-HIFU hyperthermia | 48 hours following first dose
Clearance (mL/min) of Doxil when delivered with MR-HIFU hyperthermia | 48 hours following first dose
Adverse events associated with Doxil when administered in combination with MR-HIFU hyperthermia | 6 months
Percentage of patients with relapsed or refractory solid tumors treated with MR-HIFU hyperthermia and Doxil who demonstrate disease progression at a MR-HIFU treated lesion | Through study completion, an average of 1 year
Tumor response to MR-HIFU with liposomal doxorubicin | 6 months
Percentage of patients treated with MR-HIFU hyperthermia who are able to receive hyperthermia (41-45C) to greater than 75% of the predetermined treatment volume for greater than 75% of the planned treatment duration | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center/Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903